CLINICAL TRIAL: NCT02887794
Title: Basic Auditory Processing and Acoustico-verbal Hallucinations: a Pathophysiological Study
Brief Title: Basic Auditory Processing and Auditory Hallucinations
Acronym: AUDISCHIZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-A00141-50
Record Dates: First submitted 2016-08-03; First posted 2016-09-02 (Estimated); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Schizophrenia
Keywords: pitch discrimination; auditory processing disorders; auditory perception; auditory-verbal hallucinations; theory of mind
MeSH Terms: conditions — Schizophrenia; Auditory Perceptual Disorders; Hallucinations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 30 patients with schizophrenia (Experimental): Measure the correlation between the score on the scale psychometric AHRS (Auditory Hallucination Rating Scale) to measure HAV and performance scores discrimination test psychoacoustic Tone Matching Task in subjects suffering from schizophrenia and HAV.
  Interventions: Other: Clinical and psychoacoustic measures

INTERVENTIONS:
Other: Clinical and psychoacoustic measures — Our study focuses on psychoacoustic tests, specialist care protocols (psychotherapy, neuromodulation ...) being made independently of our study, as part of medical activity of Cerletti care unit or differentiated protocols. Thus, our study shows no individual benefit for the patient. However, a better understanding of the neurophysiological mechanisms underlying auditory hallucinatory phenomenon could allow a better management of these patients in the near future

SUMMARY:
Schizophrenia is a severe psychiatric disorder that affects approximately 1% of the population worldwide. Although pathophysiology of this disease remains unclear, a growing interest is emerging for low-level sensory function, acknowledging that deficits in early stages of sensory processing are related to higher-order cognitive disturbances in schizophrenia. In the field of auditory processing, symptoms as auditory-hallucinations were found correlated with disabilities to discriminate psychoacoustic parameters of sounds.

DETAILED DESCRIPTION:
Outcomes: Our main hypothesis is that Auditory Hallucinations Rating Scale (AHRS) scores are correlated with the percentage of wrong answers in a Tone-Matching Task test. The main objective is to assess this correlation. Our other objectives are to assess correlation between AHRS as well as other symptoms scales and psychoacoustic tests assessing intensity, length discrimination of non-verbal tones and self-monitoring abilities. Impact of therapeutic procedures (neuromodulation, psychotherapy) conducted independently of our study on these psychoacoustic tests will also be assessed.

Methods: 30 subjects with schizophrenia will be included. Clinical and psychoacoustic measures will be carried out at J-0. In the case of patients receiving therapeutic procedures independently of our study, new clinical and psychoacoustic measures will be carried out at J+7 and J+30.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years old
* Meeting DSM-5.0 criteria for schizophrenia
* Auditory Hallucinations Rating Scale ≥ 8
* Negative βHCG level if woman
* Effective contraception if woman
* Consent to be included in the study

Exclusion Criteria:

* Hearing impairment
* Neurologic disorder
* Other psychiatric disorder from the DSM-5.0 section II
* Developed musical abilities (regular practice of singing or a musical instrument)
* Pregnancy
* Does not consent to be included in the study
* Lacking in legal capacity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
percentage error in discrimination test psychoacoustic Tone Matching Task | immediately after treatment
  Our main hypothesis is that Auditory Hallucinations Rating Scale (AHRS) scores are correlated with the percentage of wrong answers in a Tone-Matching Task test.

SECONDARY OUTCOMES:
Score the item hallucinations of psychometric ( positive and negative syndrome ) scale | immediately after treatment
  Rating Scale(AHRS) as well as other symptoms scales and psychoacoustic tests assessing intensity, length discrimination of non-verbal tones and self-monitoring abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Haesebaert Frédéric, PH, Principal Investigator — CH LE VINATIER
Locations (1):
- Ch Le Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No